CLINICAL TRIAL: NCT00403416
Title: 12-month Open Label, Randomized, Multicenter Study Evaluating Efficacy, Safety and Tolerability of Oral AEB071 Plus Tacrolimus (Converted to Mycophenolic Acid After 3 Months), vs. Mycophenolic Acid Plus Tacrolimus in de Novo Renal Transplant Recipients
Brief Title: Efficacy and Safety of AEB071 Plus Tacrolimus (Converted to Mycophenolic Acid After 3 Months), in Renal Transplant Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAEB071A2203
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2017-05

CONDITIONS: Kidney Transplantation
Keywords: AEB071; Tacrolimus; Mycophenolic acid; Basiliximab; Rejection; Kidney function; Immunosuppression
MeSH Terms: conditions — Rejection, Psychology | interventions — sotrastaurin; Mycophenolic Acid

ARMS (3):
- Mycophenolic Acid / tacrolimus (Active Comparator)
  Interventions: Drug: Mycophenolic Acid
- AEB071 / tacrolimus arm 1 (Experimental)
  Interventions: Drug: AEB071
- AEB071 / tacrolimus arm 2 (Experimental)
  Interventions: Drug: AEB071

INTERVENTIONS:
Drug: AEB071
  Arms: AEB071 / tacrolimus arm 1; AEB071 / tacrolimus arm 2
Drug: Mycophenolic Acid
  Arms: Mycophenolic Acid / tacrolimus

SUMMARY:
This study will evaluate the efficacy and safety of AEB071 in preventing acute rejections after kidney transplantation, when combined with tacrolimus for the first 3 months and with myfortic thereafter.

ELIGIBILITY:
Inclusion criteria

* Male and female patients of any race 18 years or older
* Adult recipients of a kidney transplant from a deceased or from a living donor
* Recipients of a functioning Kidney:. Graft must be functional no later than 36h after transplantation.

Exclusion criteria

* Need for medication prohibited by the protocol
* Patients or donors infected with hepatitis B or C, or with HIV.
* Patients with a history of cancer
* Patients with severe systemic infections Patients with heart diseases (own or family history) which are associated with an increased risk for arrhythmias.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2006-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Primary efficacy failure, defined as a composite efficacy endpoint of treated biopsy-proven acute rejection (BPAR), graft loss, death or loss to follow-up | at 6 months

SECONDARY OUTCOMES:
Renal function post-transplant Modification of diet in renal disease (MDRD) formula for Glomerular Filtration Rate) | at 6 months
Primary efficacy failure, defined as a composite efficacy endpoint of treated BPAR, graft loss, death or loss to follow-up | at 3 and 12 months
Various efficacy endpoints, using treated BPAR, treated acute rejection (AR), death, graft loss, loss to follow-up and combinations thereof. | at Month 3, 6 and 12
Changes in renal function (GFR) after replacing tacrolimus by myfortic in the AEB071 treatment arms | from Month 3 to Month 6
Safety and tolerability | at 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (28):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - University Hospitals of Cleveland, Cleveland, Ohio
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- QE II Health Sciences Center, Halifax, Canada
- France (4):
  - Hopital Kremlin Bicetre, Le Kremlin-Bicêtre
  - Hopital Hotel Dieu, Nantes
  - Hopital Necker, Paris
  - CHU de Rangueil, Toulouse
- Germany (6):
  - Universitaetsklinik Charite, Berlin
  - Klinikum der Humboldt Universitat Charite, Berlin
  - Staedt. Krankenhaus Koeln-Merheim, Cologne
  - Universitaetsklinikum Essen, Essen
  - Medizinische Hochschule Hannover, Hanover
  - Univ. - Klinikum Heidelberg, Heidelberg
- Italy (3):
  - Az. Osp. Di Bologna Polici. S. Orsola - Malpighi, Bologna
  - Azienda Opedaliera Careggi - Universita degli Studi, Florence
  - Azienda Ospedaliera di Padova - Universita degli Studi, Padua
- Spain (4):
  - Ciutat Santitaria I Univessitaria de Bellvitge, L'Hospitalet de Llobregat
  - Hospital 12 de Octubre, Madrid
  - Complejo Hospitalario Carlos Haya, Málaga
  - Hospital Doctor Peset, Valencia
- Switzerland (3):
  - Universitatsspital Basel, Basel
  - Inselspital Bern, Bern
  - Universitätsspital Zürich, Zurich
- United Kingdom (4):
  - University Hospital of Wales, Cardiff
  - Western Infirmary, Glasgow
  - Saint George's University of London, London
  - Manchester Royal Infirmary, Manchester

REFERENCES:
- See also: Results for CAEB071A2203 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2800